CLINICAL TRIAL: NCT07305649
Title: The Effectiveness of an Innovative Inhalation Training Device in Improving Medication Accuracy, Dyspnea, and Quality of Life in Elderly Patients With Chronic Obstructive Pulmonary Disease
Acronym: pMDII
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-06-003B
Record Dates: First submitted 2025-12-03; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inhaler training; pMDI; Elderly patients; Dyspnea; Quality of life; EQ-5D; CAT; mMRC; Inhaler technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel-group, two-arm randomized controlled trial design. Eligible elderly patients with COPD are randomly assigned to the control group (standard nursing guidance) or the experimental group (standard guidance plus an innovative inhaler training tool, "GoldSharp"). Outcomes are compared between groups at three time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative Inhaler Training Device (Experimental): Participants receive standard pMDI inhaler education plus training using the innovative inhalation training device (e.g., 金犀利裝置) for three sessions over two weeks.
  Interventions: Behavioral: Innovative Inhaler Training Device (金犀利); Behavioral: Standard pMDI Inhaler Education
- Standard Nursing Education (Active Comparator): Participants receive standard pMDI inhaler education only, based on established clinical nursing guidelines. No additional device or interactive training is provided. The education includes written and verbal instructions on proper pMDI use.
  Interventions: Behavioral: Standard pMDI Inhaler Education

INTERVENTIONS:
Behavioral: Innovative Inhaler Training Device (金犀利) — This intervention involves the use of an innovative inhaler training device designed to assist elderly COPD patients in mastering the correct pMDI inhalation technique. The device provides visual and auditory feedback during training and is used in conjunction with individualized nursing instruction. The goal is to improve medication administration accuracy, reduce dyspnea, and enhance quality of life.
  Arms: Innovative Inhaler Training Device
Behavioral: Standard pMDI Inhaler Education — Participants receive standard pMDI inhaler education only, based on established clinical nursing guidelines. No additional device or interactive training is provided. The education includes written and verbal instructions on proper pMDI use.

SUMMARY:
This study aims to evaluate the effectiveness of an innovative inhaler training device, "Golden Rhino" (pMDI Practice Tool), in improving inhalation technique accuracy, dyspnea severity, and quality of life among elderly patients with chronic obstructive pulmonary disease (COPD). The device integrates a weighted valve and musical cues to guide patients in synchronizing their breath with proper pMDI inhalation technique. Participants will be randomly assigned to either standard nursing guidance or nursing guidance plus device-based training. Outcome measures include pMDI usage accuracy, dyspnea severity, and EQ-5D quality of life scores at baseline and follow-up.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) remains a leading cause of morbidity among older adults. Effective pMDI inhalation technique is critical for symptom control, yet improper use is common among elderly patients, especially those with cognitive decline or low health literacy. To address this, we developed an innovative training tool, "Golden Rhino" (patent number M647974, Taiwan), which utilizes a weight-calculated valve to simulate proper inhalation flow (20-60 L/min) and incorporates music cues to assist in breath timing (inhale, hold, exhale).

This randomized controlled trial investigates whether adding this tool to routine nursing education improves pMDI technique accuracy, alleviates dyspnea (via mMRC and CAT), and enhances quality of life (via EQ-5D-5L) in elderly COPD patients. Eligible participants aged 65 years and above will be enrolled from a medical center. Intervention group patients will use the device under nursing instruction for one week. The control group will receive standard verbal instructions only. Assessments occur at baseline, one week, and one month post-intervention.

The device is a non-commercial, research-use-only prototype with no financial gain or commercialization involved. This study has disclosed all relevant intellectual property in the IRB process and participant consent forms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Clinically diagnosed with Chronic Obstructive Pulmonary Disease (COPD) according to GOLD criteria
* Currently using pressurized Metered Dose Inhaler (pMDI) medications
* Ability to communicate and understand instructions in Mandarin or Taiwanese
* Willing to participate and provide informed consent

Exclusion Criteria:

* Diagnosis of severe cognitive impairment (e.g., dementia) that may interfere with participation
* Acute COPD exacerbation requiring hospitalization within the past 30 days
* Concurrent enrollment in another interventional clinical trial
* Severe visual or hearing impairment that may limit the ability to follow inhaler training instructions
* Other diagnosed pulmonary diseases (e.g., lung cancer, pulmonary fibrosis) that may affect the assessment of COPD outcomes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in dyspnea severity | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  Dyspnea severity will be measured using the modified Medical Research Council (mMRC) dyspnea scale. The mMRC is a 5-point scale ranging from 0 (no dyspnea) to 4 (dyspnea on minimal exertion). Participants will self-report their score at baseline, post-intervention, and 4-week follow-up. Reduction of at least 1 point is considered clinically significant.
Correct use of pMDI inhaler | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  Correct inhaler technique will be assessed using a 10-item standardized checklist. Each item is scored as correct (1) or incorrect (0). Total scores range from 0 to 10. Participants will be observed by trained nursing staff during inhaler use at three time points: baseline, post-intervention (2 weeks), and follow-up (4 weeks). A score ≥9 is considered correct use.
Health-related quality of life (HRQoL) | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  Health-related quality of life will be assessed using the EQ-5D-5L instrument, including both the index score (calculated using the China value set from Luo et al., 2017, DOI: 10.1007/s10198-017-0870-1
  ) and the EQ-VAS score. The EQ-5D index score ranges from <0 (worse than death) to 1 (perfect health). The EQ-VAS is a visual analog scale from 0 to 100 representing self-rated health

SECONDARY OUTCOMES:
Change in peak expiratory flow (PEF) | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  Peak expiratory flow will be measured using the MIR Smart One digital spirometer. Participants will perform three trials, and the highest value will be recorded in liters per minute (L/min). PEF reflects airway obstruction and inhalation-exhalation efficacy. Measurements will be taken at baseline, post-intervention (2 weeks), and follow-up (4 weeks).
Change in forced expiratory volume in one second (FEV₁) | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  FEV₁ will also be assessed using the MIR Smart One device. Three measurements will be taken, and the highest value recorded in liters (L). FEV₁ is a standard measure of lung function in COPD and will be compared across time points to assess improvement.
Change in COPD Assessment Test (CAT) score | Pre-intervention, immediately post-intervention, 4 weeks, 12 weeks
  The CAT is an 8-item self-administered questionnaire assessing the impact of COPD on health status. Each item is scored from 0 to 5, with a total score range of 0-40. Higher scores indicate worse health status. A reduction of 2 or more points is considered clinically meaningful.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided